CLINICAL TRIAL: NCT03572179
Title: Evaluation of Fixed Mandibular Retainer Using 3D Printed Positioning Tray Versus Direct Bonding Technique A Randomized Clinical Trial
Brief Title: Evaluation of Fixed Mandibular Retainer Using 3D Printed Positioning Tray Versus Direct Bonding Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raghda Alaa (Other)
Responsible Party: Sponsor-Investigator, Raghda Alaa, principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CEBD-CU-2018-04-28
Record Dates: First submitted 2018-06-09; First posted 2018-06-28 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Orthodontic Appliance Complication
Keywords: 3d printed positioning tray

STUDY DESIGN:
Intervention Model Description: all patient will receive a modified indirect technique for bonding fixed mandibular retainer and the key of modification is the fabrication of 3D printed digital positioning tray for placement of retainer with holes for composite pads for its direct application using 3 shape Ortho analyser Software ® instead of conventional indirect retainer fabrication method
Who Masked: Outcomes Assessor
Masking Description: Participants Patients can detect the transfer tray so blinding is not possible Operator The main operator is responsible for the bonding so the blinding is not possible Assessor The assessor (different from main operator will carry out the measurement blindly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): After finishing orthodontic treatment, all patient will receive a modified indirect technique for bonding fixed mandibular retainer and the key of modification is the fabrication of 3D printed digital positioning tray for placement of retainer with holes for composite pads for its direct application using 3 shape Ortho analyser Software ® instead of conventional indirect retainer fabrication method
  Interventions: Device: 3d printed positioning tray
- Control Group (No Intervention): All patients of this group will follow conventional steps of direct bonding procedure of fixed mandibular retainer

INTERVENTIONS:
Device: 3d printed positioning tray — 3d printed positioning tray for lingual fixed retainer placement in treatment group
  Arms: Treatment Group

SUMMARY:
Although there are many studies in the literature concerning methods of bonding of mandibular retainers whether directly or indirectly, there is a very limited evidence regarding their chair side time and bond failure. Also there are scarce data on fixed mandibular retainers bonded using 3D printed positioning tray.Thus, conducting a well-designed randomized clinical trial evaluating the chair side time and bond failure of 3d printed positioning tray and direct bonding method of fixed mandibular retainer.Null hypothesis is thatThe time needed for direct indirect bonding using 3D digital positioning tray of a mandibular fixed retainer is shorter than the time needed for direct bonding, and there is no difference in failures between the 2 bonding methods

DETAILED DESCRIPTION:
Statement of the problem:

- Although there are many studies in the literature concerning methods of bonding of mandibular retainers whether directly or indirectly, there is a very limited evidence regarding their chair side time and bond failure. Also there are scarce data on fixed mandibular retainers bonded using 3D printed positioning tray.

Choice of the comparator:

In the ongoing study, direct bonding of mandibular fixed retainer will be the control group. Thus, conducting a well-designed randomized clinical trial evaluating the chair side time and bond failure of 3d printed positioning tray and direct bonding method of fixed mandibular retainer.

Study rationale:

To evaluate and compare bond failure and chair side time by 3D printed positioning tray and direct bonding method of mandibular fixed retainer.

Null hypothesis:

1. The time needed for direct indirect bonding using 3D digital positioning tray of a mandibular fixed retainer is shorter than the time needed for direct bonding, and (2) there is no difference in failures between the 2 bonding methods.

   Research question:

   Will the 3D digital positioning tray reduce chair side time, bond failure during retainer placement in patient with need of fixed bonded mandibular retainer, when compared to direct bonding method?

   Aim of the study:

   To evaluate chair side time and bond failure of 3D digital positioning tray during mandibular retainer placement and direct bonding of mandibular retainer.
2. Objectives

   Primary objective To evaluate effect of 3D Digital positioning Tray on chair side time Secondary outcome Immediate bond failure and bond failure during first 6 month of placement of mandibular fixed retainer.

   PICOTs format:

   P: patient with the need of fixed bonded mandibular retainer after orthodontic treatment I: 3D printed Digital positioning Tray for bonding mandibular retainer. C: conventional direct bonding of mandibular retainer O: chair side time, immediate bond failure and bond failure during first 6 month.

   Outcome Name,Measuring Tool and Measuring unit Primary is the Chair side Time measured by Digital stopwatch in Seconds Immediate Bond Failure is the Number of Debonded mandibular fixed retainer measured in Numerical value Bond failure during first 6 month follow up by the Number of Debonded mandibular fixed retainer measured in Numerical value

   T: Immediate and T2: 6 month follow up S: Randomized controlled trial.
3. Trial Design This trial is designed as a parallel, randomized, controlled trial with allocation ratio 1:1.It will be performed at the educational hospital of the Faculty of Oral & Dental Medicine, Cairo University.

Materials & Methods:

I. Participants, Intervention and Outcomes

A) Study setting:

* Source of patients: patients who finished their orthodontic treatment at the outpatient clinic in Orthodontic department, Faculty of Oral and Dental Medicine, Cairo University, Cairo government, Egypt.
* Time: 2017-2018 The study will last for 6 months.

C) Intervention Treatment Group After finishing orthodontic treatment, all patient will receive a modified indirect technique for bonding fixed mandibular retainer and the key of modification is the fabrication of 3D printed digital positioning tray for placement of retainer with holes for composite pads for its direct application using 3 shape Ortho analyser Software ® instead of conventional indirect retainer fabrication method The sample selection and screening for inclusion of patients in clinical trial will be performed at all patients at clinic of Orthodontic department, Faculty of Oral and Dental Medicine, Cairo University.

Scanning of impression and designing the digital tray Lower impression is taken for each patient and the cast will be carefully scanned by desktop laser scanner for production of digital cast, using 3 shape ortho analyser Software®, the tray will be designed Fabrication and printing of the digital tray Using Dent1 3D printer® (Mogassam®, Greek campus, Cairo, Egypt), the tray will be printed Clinical application of the digital tray

* Teeth to be bonded are polished and etched.
* Teeth isolation & moisture control are achieved.
* Dead Soft Stainless Steel wire is placed and adapted in its place in the digital tray.
* Placement of the tray in the patient mouth on the prepared teeth
* Adhesive bond is applied to teeth and then curing of the adhesive bonding.
* 3M ® composite (3M Unitek company , Monrovia, California, USA) is placed in the printed tray holes and any excess composite will be removed and then light curing is done.
* Time will be recorded during this step

Removal of digital tray After insuring complete curing of the composite the digital tray is then removed from patient mouth, Bond failure of composite pads will be checked in this step and recorded.

Control Group All patients of this group will follow conventional steps of direct bonding procedure of fixed mandibular retainer

* Pumice and polish the lingual surface of teeth on which retainer is to be bonded
* The retainer wire is prefabricated by incorporating perpendicular pieces of 1.5"-2" ligature wire at interdental region of respective teeth
* The retainer wire is then adapted on the tooth surface. The short ligatures are passed interdentally one occlusal to contact point and other gingival to contact point and tied over.
* Bonding procedure after etching and application of sealant is carried out.
* Enough adhesive should be used. Light curing is done.
* 3M ® composite (3M Unitek company, Monrovia, California, USA) is placed then light curing is done.
* Cut the ligature wires and pull them laically to disengage.
* Time will be recorded during this step

F) Sample Size calculation:

the sample is increased to a total size of 20 participants; 10 in each arm.

G) Recruitment strategy:

* Patients will be selected from the outpatient clinic of the orthodontic Department - Cairo University
* Consecutive sampling is done through screening of patients. This will continue until the target population is achieved.
* Identifying and recruiting potential subjects is achieved through patient database.

II. Assignment of Interventions

A) Sequence generation:

It will be performed as 1:1 allocation. The sequence of the two groups will be done by computer generated random numbers. This will be done by using Microsoft Office Excel 2013 sheet

B) Allocation Concealment:

Random numbers obtained by random sequence generation will be written on white papers, each paper will be kept in sealed envelope. Sealed envelopes will be kept in box at the secretary of orthodontic department office.

C) Implementation:

Implementation will be carried out in the secretary of the orthodontic department at the Faculty of Oral and Dental Medicine, Cairo University.

D) Blinding:

Participants Patients can detect the transfer tray so blinding is not possible Operator The main operator is responsible for the bonding so the blinding is not possible Assessor The assessor (different from main operator will carry out the measurement blindly

ELIGIBILITY:
Inclusion Criteria:

* • Patients with properly finished orthodontic treatment according to ABO standards.

  * the presence of the 4 mandibular incisors and the 2 mandibular canines,
  * No active caries, restorations, fractures, or periodontal disease of these teeth
  * Patient with Good oral hygiene

Exclusion Criteria:

* • Patients with no need of fixed bonded mandibular retainer

  * No or poor patient's co operation
  * Abnormal morphology of anterior teeth
  * Bad oral hygiene

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
chairside time | follow up up to 6 month
  chairside time for bonding fixed lingual mandibular retainer using stopwatch in measured seconds

SECONDARY OUTCOMES:
bond failure | 6 month follow up
  bond failure of composite per tooth measuered in numerical value

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No